CLINICAL TRIAL: NCT04212312
Title: Repeat Versus Single Course of Betamethasone in Twin Pregnancies
Brief Title: Single Versus Repeat Betamethasone in Twin Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yaniv Zipori MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0484-19
Record Dates: First submitted 2019-11-02; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Twin; Complicating Pregnancy
Keywords: Betamethasone; Twin pregnancy; Repeat course; Single course
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single course of Betamethasone: Women with twin pregnancy who received 1 course of betamethasone between 24 - 34 weeks' gestation.
- Repeat course of Betamethasone: Women with twin pregnancy who received 2 courses (Repeat course) of betamethasone between 24 - 34 weeks' gestation.

SUMMARY:
Thus far no robust data exist as to the effect of repeted course of antenatal corticosteroids in twin pregnancies. The investigators hypothesized that repeat course of betamethasone would further reduce neonatal morbidity in twins born before 34 weeks' gestation when compared with single dose.

DETAILED DESCRIPTION:
Observational data suggest benefits in multiple gestations exposed to antenatal corticosteroids, although these studies have not consistently reported a statistical benefit or the benefits achieved in singletons. Nevertheless, based on the improved outcomes reported in singleton gestations, one course of antenatal corticosteroids is administered to all patients who are between 24 weeks and 34 weeks of gestation and at risk of delivery within 7 days, irrespective of the fetal number. Moreover, "a repeat course" of antenatal corticosteroids should also be considered in women who are less than 34 weeks of gestation who have an imminent risk of preterm delivery within the next 7 days, and whose prior course of antenatal corticosteroids was administered more than 14 days previously, again, irrespective of the fetal number.

The objective of the current study is to evaluate fetal outcomes in twin pregnancies following repeat betamethasone administration during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Study group - women who received 2 courses of betamethasone between 24 - 34 weeks' gestation.
* Control comparison group - women who received 1 course of betamethasone between 24 - 34 weeks' gestation.

Exclusion Criteria:

* singletone pregnancies
* higher order multiple pregnancies (triplets and above)
* known major congenital anomaly

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women with twin pregnancies, and who received Betamethsone during the course of their pregnancy for threatened preterm labor.
Study Population: Pregnant women carrying twins, and who received antenatal Betamethasone between 24-34 weeks' gestation for threatened preterm labor.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of respiratory morbidity after single versus repeat course of betamethasone for threatened preterm labor between 24-34 weeks' gestation | 1 year
  The incidence of respiratory morbidity after single versus repeat course of betamethasone for threatened preterm labor between 24-34 weeks' gestation

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Zipori, M.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet, maybe in the future or part of a meta-analysis